CLINICAL TRIAL: NCT01583998
Title: Electronic-Measurement Based Care (e-MBC) for Major Depressive Disorder (MDD)
Brief Title: Electronic-Measurement Based Care for Major Depressive Disorder
Acronym: e-MBC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: UTSW Family Medicine refused to comply with agreement to implement study after department head left university. Attempts to implement elsewhere failed.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, David W. Morris, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R03MH092509-01 (NIH)
Record Dates: First submitted 2012-04-19; First posted 2012-04-24 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; MDD; Depression; Measurement Based Care; MBC; electronic health records; EHR; electronic medical records; EMR
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- e-MBC (Active Comparator): Patients will receive e-MBC
  Interventions: Behavioral: e-MBC
- Treatment as Usual Control (No Intervention): Patients receive standard treatment

INTERVENTIONS:
Behavioral: e-MBC — antidepressant treatment
  Other Names: e-MBC for MDD
  Arms: e-MBC

SUMMARY:
The pilot study will evaluate whether electronic-Measurement Based Care (e-MBC) using the UT Southwestern MyChart personal health record is feasible, associated with patient and health care team satisfaction, and improves treatment outcomes compared to a standard treatment model. The project will be conducted in the Simmons Cancer Center Clinic at the University of Texas Southwestern Medical Center, Dallas as a collaborative effort between the Departments of Psychiatry, Oncology, and Family and Community Medicine. The primary patient population will include adults with significant depression and/or starting an antidepressant treatment and/or experiencing a treatment change. The study will compare two groups, an e-MBC group and an office-based standard care MBC group. Study staff will explain the study to the patients, specifically explaining that study participants will receive either office-based MBC or e-MBC. Eligible participants must be willing to receive either form of treatment monitoring. Participating patients will be randomly assigned to receive either e-MBC or office-based MBC. In the e-MBC group once a month the study nurse will send a prompt from the participating patients treating physician requesting the patient to use the MyChart system to fill-out the MBC scales. Beyond these monthly assessments, patients will be encouraged to utilize the MyChart MBC assessments (e-MBC) at any time to communicate with their physician. Patients experiencing difficulties using the e-MBC system will be given additional instruction by the study nurse. Patients and physicians will be trained in the use of the eMBC system. In the office-based MBC group the study nurse will schedule monthly treatment visits and request the patient call as needed to report symptoms. The evaluation period will be 6 months.

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) is a serious, debilitating illness that affects persons of all ages, races, and socioeconomic backgrounds. Despite the availability of new and effective treatments over the last 20 years, recent evidence continues to demonstrate high rates of inadequate antidepressant medication treatment in practice settings. Practitioners vary widely in how they assess treatment outcomes, including symptoms, function, side-effect frequency and burden. In contrast to other chronic medical conditions such as diabetes mellitus, back/neck problems, or hypertension, clinicians treating patients with depression do not routinely evaluate measurement-based care (MBC) treatment parameters. MBC provides an essential framework for physicians to approach depression treatment consistent with their approach for other common disorders. MBC is an effective means to provide patient-centered care for MDD, personalizing treatment decisions based on patient progress and their ability to tolerate the medication.

A key barrier to patient adherence with MBC treatment is that the approach requires patients to return to the clinic for several follow-up visits. The necessity of treatment visits varies widely among patients. Thus far, physicians using MBC for the treatment of MDD do not have a complete set of tools that are practical to use and allow treatment to be truly personalized patient-centered care.

One solution to this problem is to use an enhanced electronic personal health record, such as the MyChart system. This system could be easily modified to include the central elements of MBC for depression to allow for the systematic assessment of a patient's depressive symptom severity, antidepressant tolerability, and adherence to treatment in a timely fashion. This information would be available to allow the physician to provide patient-centered care by utilizing standardized assessment to personalize treatment for depression. The proposed electronic-MBC (e-MBC) addresses a critical gap in depression treatment by providing regularly-scheduled drug monitoring and continuity of care, in the face of limited patient and clinic resources.

Information technology (IT) systems have been effectively integrated into the medical treatment of patients but have yet to have substantial impact at the point-of-care. Applying e-MBC methods allows physicians to utilize existing information technology systems to improve depression treatment at the point-of-care. The key features of the proposed e-MBC approach are that it can be seamlessly integrated into standard clinical practice, and requires no additional IT knowledge or training to be effectively utilized by physicians and clinical staff.

In this pilot study the investigators will compare standard treatment (office based antidepressant management) to a group receiving scheduled electronic MBC assessments via an enhanced personal health record system (e-MBC). To date, no one has published feasibility studies evaluating the use of personal health records for measurement-based care of depression patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must plan to continue living in the clinic area throughout the study
* Patients must be 18 to 65 years of age
* Patients must give written informed consent
* Patient must have clinically significant depression and/or starting an antidepressant treatment and/or experiencing a antidepressant treatment change
* Patients must be willing and able to use MyChart to communicate with their physician

Exclusion Criteria:

* Patients with a current Axis I diagnosis of Bipolar disorder or Schizophrenia
* Patients who cannot read and understand English since all research instruments are not yet translated and validated in Spanish or other languages
* Patients whose clinical status requires inpatient treatment at the time of baseline interview.
* Current substance abuse or dependence
* Patients with current suicidal ideation
* Patients with general medical conditions that contraindicate antidepressant medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Every 30 days for 6 months
  Depression severity assessment

SECONDARY OUTCOMES:
Frequency, Intensity, and Burden of Side Effect Rating (FIBSER) | Every 30 days for 6 months
  Antidepressant side effects
Patient Satisfaction Questionnaire (PSQ) | At the end of study treament (6 months from the first assessment)
  Assesses satisfaction with care
Physician Evaluation of Ease of Use Survey (EEUS) | At the end of study treament (6 months from the first assessment)
  Physicians' perception of the ease of use of the e-MBC system
Physician Evaluation of Usefulness Survey (EUS) | At the end of study treament (6 months from the first assessment)
  Physicians' perception of the usefulness of the e-MBC system

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas Southwestern Medical Center, Dallas, Texas, United States